CLINICAL TRIAL: NCT00483834
Title: A Phase II Study of Bevacizumab, Irinotecan and Capecitabine in Patients With Previously Untreated Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XELIRI-A
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Cancer
Keywords: Bevacizumab; Avastin; CPT-11; Irinotecan; Camptothecin-11; Capecitabine; Xeloda; Metastatic; Colorectal; Colon; Rectal
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Bevacizumab; Vascular Endothelial Growth Factor A; Irinotecan; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab, Irinotecan and Capecitabine (Experimental): Evaluate the efficacy and toxicity of bevacizumab, irinotecan and capecitabine as first-line treatment for patients with metastatic colorectal cancer
  Interventions: Drug: Bevacizumab; Drug: Irinotecan; Drug: Capecitabine

INTERVENTIONS:
Drug: Bevacizumab — 7.5mg/kg, IV, day 1 of each cycle
  Other Names: Avastin; VEGF; rhuMAb
Drug: Irinotecan — 200mg/m^2, IV, day 1 each cycle
  Other Names: CPT-11; hydrochloride trihydrate; Camptosar
Drug: Capecitabine — 1000mg/m^2 or 750mg/m^2 for patients over 65yrs old PO BID, day 1-14 each cycle
  Other Names: Xeloda

SUMMARY:
Bevacizumab has recently been shown to improve survival when combined with chemotherapy in patients with previously untreated metastatic colorectal cancer. Bevacizumab is usually given together with infusional 5-FU, which requires a central line. A central line is inconvenient for patients, and may increase risk of infection, and thrombosis. Furthermore, a central line increases resource demands for interventional radiology, chemo daycare. Capecitabine is administered orally, and converted to 5-FU intracellularly. Chronic administration of capecitabine mimics infusional 5-FU. This study is designed to evaluate whether the combination of irinotecan, capecitabine and bevacizumab is effective as a first-line therapy for patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
The FOLFIRI regimen has become the standard 1st line therapy for metastatic colorectal cancer in Canada. This regimen consists of irinotecan in combination with bolus 5-FU/leucovorin, followed by 46-hour infusional 5-FU every 2 weeks. It requires a central line and an infusion pump for delivering 5-FU, and necessitates at least 2 visits to the chemotherapy units every 2 weeks, which not only incurs additional cost and inconvenience to patients, but also increases the risk of complications such as thrombosis and infection due to the central line. In addition, due to resources limitations, patients often have to wait several weeks for central line placement. The XELIRI (irinotecan and capecitabine) regimen has been in use at the Princess Margaret Hospital (PMH) as the first-line treatment of patients with metastatic colorectal cancer since May, 2003. The choice of XELIRI over FOLFIRI was made in efforts to reduce demands on resources, enable patients to start therapy sooner, increase patient convenience and potentially reduce complications associated with central venous access. The regimen consists of irinotecan 250 mg/m2 IV on day 1 and capecitabine 1000 mg/m2 PO BID from days 1-14 every 3 weeks. The dose was reduced to irinotecan 200 mg/m2 on day 1 and capecitabine 750 mg/m2 in patients > 65 years old or in patients with renal impairment. So far, 101 patients have been treated on this regimen at PMH. Among 76 patients evaluable for response, there have been 34 confirmed partial responses (44.7%) and a further 18 patients with stable disease (23.7%), for a disease control rate of 68.4%. Furthermore, this regimen was well tolerated with main side effects being diarrhea and neutropenia. With availability of bevacizumab, 12 patients were treated with the XELIRI regimen in combination with bevacizumab at PMH as part of the BEAT (Bevcizumab Expanded Access Trial ) study up to October, 2005. Of 10 patients who were treated with 3 or more cycles of chemotherapy, there were 7 confirmed partial responses and 2 additional patients with stable disease. One patient with non-measurable but evaluable disease had marked reduction in infiltration in the sacrum. There were no instances of GI perforation, febrile neutropenia, or toxic death. The median number of cycles of treatment was 6, and 9 of 12 patients are still receiving treatment. There were, however, a total of 8 dose reductions of capecitabine in 6 patients, with majority of dose reductions as a result of hand-foot syndrome. Although these efficacy and toxicity data are extremely encouraging, the small number of patients limits the potential application of these data.Because of the encouraging preliminary results, it is necessary to conduct a prospective clinical study to further evaluate the efficacy and toxicity of irinotecan, capecitabine and bevacizumab combination (the XELIRI-A regimen) as first-line chemotherapy for patients with advanced colorectal cancer. Results from this study would provide the scientific basis for a randomized phase III study to compare the XELIRI-A regimen to the IFL (FOLFIRI) + bevacizumab regimen. Furthermore, it will have practical implications for our centre. Compared to infusional or bolus 5-FU based regimens, the XELIRI-A regimen will reduce workload in the chemotherapy daycare unit and drug costs, reduce demands for resources such as infusion pumps and interventional radiology time, enable patients to start therapy sooner, and improve patient convenience.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed colorectal cancer which is recurrent or metastatic, and not amendable to surgical resection or radiation.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan. See section 11.2 for the evaluation of measurable disease.
* Patients must have had no previous chemotherapy or treatment with an investigational agent for recurrent or metastatic disease. Prior chemotherapy in the adjuvant setting for colorectal cancer is acceptable. Prior surgery or radiotherapy for recurrent or metastatic disease is acceptable, however, patients must be adequately recovered from the effects of these treatments. At least 6 weeks must have elapsed from major surgery and 4 weeks must have elapsed from any radiation therapy.
* Age >18 years. Because no dosing or adverse event data are currently available on the use of bevacizumab in combination with capecitabine and irinotecan in patients <18 years of age, children are excluded from this study.
* Estimated life expectancy of greater than 3 months.
* ECOG performance status 0, 1, or 2 (or Karnofsky >60%; see Appendix A).
* Patients must have normal organ and marrow function as defined below:

leukocytes >/= 3,000/mcL absolute neutrophil count >/= 1,500/mcL platelets >/= 100,000/mcL hemoglobin >/= 90 g/L total bilirubin </= 1.5 x upper limit of normal AST(SGOT)/ALT(SGPT) </= 2.5 x upper limit of normal creatinine within normal institutional limits OR creatinine clearance >/= 50 mL/min/1.73 m2 for patients with creatinine levels above institutional normal proteinuria < 2+ on dipstick patients with >/= 2+ proteinuria on urine dipstick at baseline should undergo a 24-hour urine collection, and must have </= 1g protein / 24 hours

* Appropriate imaging investigations, including chest X-rays and / or CT/MRI of chest / abdomen / pelvis or other scans as clinically indicated to document all sites of disease must be performed within 28 days of study entry.
* The effects of bevacizumab on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because antiangiogenic agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study and for a period of four weeks after cessation of study therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid malignancies curatively treated with no evidence of disease for ≥ 5 years.
* Patients may not be receiving any other investigational agents.
* Patients with known metastases in the central nervous system.
* Any condition that does not permit compliance with the study protocol
* Previous history of gastrointestinal perforation, uncontrolled gastrointestinal bleeding, uncontrolled thromboembolism
* Presence of uncontrolled hypertension and / or proteinuria. Patients must have systolic blood pressure ≤ 150 mmHg and diastolic blood pressure ≤ 100 mmHg, and be on stable blood pressure medication at the time of study entry. Patients discovered to have ≥ 1+ proteinuria at baseline, should undergo a 24-hour urine collection and must have < 500 mg of protein / 24 hours.
* History of allergic reactions, or intolerance, attributed to compounds of similar chemical or biologic composition to 5-fluorouracil, irinotecan, or bevacizumab.
* Women who are pregnant or breastfeeding are excluded from this study because bevacizumab is an antiangiogenic agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with bevacizumab, breastfeeding should be discontinued if the mother is treated with bevacizumab. These potential risks may also apply to other agents used in this study.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with the agents used in this study. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Patients with active cardiovascular disease, i.e., unstable angina, New York Heart Association grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medications, or grade II or greater peripheral vascular disease. In addition, patients with arterial thrombosis, myocardial infarction, and cerebral vascular accidents (stroke / transient ischemic attach (TIA)) within 6 months prior to study entry will be excluded.
* Patients who had major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to the first study treatment, or anticipation of need for major surgical procedure during the course of the study; minor surgical procedures within 7 days prior to study treatment start.
* Planned radiotherapy for underlying disease.
* Serious non-healing wound or ulcer.
* Evidence of bleeding diathesis or coagulopathy.
* Current or recent (within 10 days prior to study treatment start) use of full dose oral or intravenous anticoagulants or thrombolytic agents. Patients on low molecular weight heparins are allowed to participate in the study. Patients with anticoagulation for maintenance of patency of permanent indwelling intravenous catheters will be eligible. However, INR should be monitored closely if patients are taking low-dose coumadin for this purpose.
* Ongoing treatment with aspirin ( > 325 mg/day) or other medications known to predispose to gastrointestinal ulceration.
* Patients who have received prior radiation therapy to > 15% of bone marrow (see Appendix D), or standard pelvic radiation for rectal cancer.
* Patients with predisposing colonic or small bowel disorders in which symptoms are uncontrolled as indicated by pre-treatment/baseline pattern of > 3 loose stools daily in patients without a colostomy or ileostomy. Patients with a colostomy or ileostomy may be entered as the investigator's discretion.
* Patients with partial or complete bowel obstruction, known chronic malabsorption, total colectomy or other major abdominal surgery that might result in substantial alteration in absorption of oral medications.
* Patients with known Gilbert's syndrome.
* Patients who were started on phenytoid, phenobarbital, carbamazepine or any other enzyme-inducing anti-convulsant drug (EIACD) within 7 days prior to the first study treatment or patients who are unable or unwilling to discontinue EIACD use or switch to a non-EIACD at least 7 days prior to the first study treatment. Concomitant use of gabapentin or other non-EIACDs is permitted.
* Patients who are unable or unwilling to discontinue St. John's wort (hypericum perforatum) at least 14 days prior to the first study treatment; Patients who are taking fluconazole / ketoconazole at the time of first study treatment.
* Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication.
* Organ allografts requiring immunosuppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | Radiological evaluation every 9 weeks, with confirmatory scans 4 weeks after objective response
  To determine the objective response rate (ie. the rate of partial response plus complete response as defined by RECIST criteria) of irinotecan, capecitabine and bevacizumab (XELIRI-A) in patients with previously untreated metastatic colorectal cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Chen, Principal Investigator — Princess Margaret Hospital, University Health Network
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Renouf DJ, Welch S, Moore MJ, Krzyzanowska MK, Knox J, Feld R, Liu G, MacKay H, Petronis J, Wang L, Chen E. A phase II study of capecitabine, irinotecan, and bevacizumab in patients with previously untreated metastatic colorectal cancer. Cancer Chemother Pharmacol. 2012 May;69(5):1339-44. doi: 10.1007/s00280-012-1843-9. Epub 2012 Feb 15. PMID 22349811